CLINICAL TRIAL: NCT02298413
Title: Clinical Study on Absorb Polylactic, Reabsorbable Coronary Scaffold (RAI)
Brief Title: Italian Absorb Registry
Acronym: BVS-RAI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Collaborators: Fatebenefratelli and Ophthalmic Hospital (Other); Bolognini Hospital (Unknown); Ospedale Regionale di Aosta (Unknown); Ospedali Riuniti di Ancona (Unknown); S. Giacomo Hospital (Other); Azienda U.L.S.S n.9 Ospedale di Treviso Ca Foncello (Unknown); Ospedale San Bortolo di Vicenza (Other); Azienda Ospedaliera Brotzu (Other); San Giuseppe Moscati Hospital (Other); Azienda Sanitaria Locale USL 13 Ospedale Mazzoni di Ascoli Piceno (Unknown); S. Andrea Hospital (Other); Ospedale Monaldi di Napoli (Unknown); Azienda Ospedaliera di Padova (Other); Ospedale della Misericordia di Grosseto (Unknown); Ospedale Santa Corona di Pietra Ligure (Unknown); Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Principal Investigator, Dr Giuseppe Steffenino, MD, Ospedale Santa Croce-Carle Cuneo
Other Study IDs: RAI-Registro Absorb Italiano
Record Dates: First submitted 2014-11-15; First posted 2014-11-24 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: PCI with Absorb scaffold — Implantation of biovascular scaffold during PCI
  Other Names: biovascular resorbable scaffold

SUMMARY:
The investigators aim at evaluating the long-term (5-year) clinical outcome following Absorb BVS implantation in a real world, all-comers population of consecutive patients, as treated according to the indications, techniques and protocols used in the participating institutions.

DETAILED DESCRIPTION:
Long-term data after implantation of coronary BVS is scarce, especially in subgroups of patients with diabetes or chronic kidney disease, and in those with complex coronary lesions and/or multivessel disease.

Although the use of BVS is very promising in younger patients with one or more of the above characteristics, evidence of benefit is not available.

The BVS-RAI Registry is a spontaneous initiative of a group of Italian interventional cardiologists who are interested in assessing the results of their interventional practice with BVS, by sharing data.

The BVS-RAI Registry has been created in joint-venture with Centro di Ricerche Farmacologiche e Biomediche "Mario Negri Sud", and is not recipient of funding or benefits originating from the BVS manufacturer or seller. BVS devices are regularly purchased by the participating centres.

Each participating centre is willing to input data of all consecutive patients treated with BVS, with a minimum of 50, and to report on follow-up for at least 5 years. Patient recruitment is not directed per protocol, nor is it rewarded. Patients who give informed consent are included in the BVS-RAI Registry after BVS implant has been performed following the indications, techniques and protocols used in each of the participating institutions.

Baseline patient clinical data, with special attention to biochemistry and drug treatment in patients with diabetes and CKD, as well as angiographic and intravascular imaging data are entered into a web-based Case Report Form.

Follow-up data from outpatient visits or phone interviews, subsequent admissions and coronary angiograms following the protocols being used in each of the participating institutions are prospectively collected and entered into the database.

All data in the CRF is visible to all registered participants at all times. Endpoints are: target lesion and target vessel failure, BVS thrombosis, new revascularisation, myocardial infarction and death. Documentation of those events is required for adjudication by an independent committee.

ELIGIBILITY:
Inclusion Criteria:

* Successful implantation of 1 or more coronary BVS
* Age <75 years
* Patient's informed consent

Exclusion Criteria:

* None

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is an all-comers study, and includes all consecutive patients who have been treated with 1 or more BVS in the study time lapse in each participating centre
Sampling Method: Non-Probability Sample
Enrollment: 1520 (Actual)
Dates: Start 2013-05; Primary Completion 2016-11 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Scaffold thrombosis | 1 year
  acute, subacute, late and very late
Target lesion revascularization | 1 year
  ischemia or angiographic-driven

SECONDARY OUTCOMES:
MACE | 5 year
  Cardiac death, TLR, myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Ielasi, MD, Principal Investigator — AO Seriate; Bernardo Cortese, MD, Principal Investigator — AO Fatebenefratelli; Donatella Corrado, PhD, Principal Investigator — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- SSD Emodinamica Dip Cardiovasc ASO S.Croce, Cuneo, Italy

REFERENCES:
- [Derived] Cortese B, Ielasi A, Moscarella E, Loi B, Tarantini G, Pisano F, Durante A, Pasquetto G, Colombo A, Tumminello G, Moretti L, Calabro P, Mazzarotto P, Varricchio A, Tespili M, Latini RA, Defilippi G, Corrado D, Steffenino G; RAI Investigators. Thirty-Day Outcomes After Unrestricted Implantation of Bioresorbable Vascular Scaffold (from the Prospective RAI Registry). Am J Cardiol. 2017 Jun 15;119(12):1924-1930. doi: 10.1016/j.amjcard.2017.03.017. Epub 2017 Mar 29. PMID 28438304
- [Derived] Cortese B, Ielasi A, Varricchio A, Tarantini G, LaVecchia L, Pisano F, Facchin M, Gistri R, D'Urbano M, Lucci V, Loi B, Tumminello G, Colombo A, Limbruno U, Nicolino A, Calzolari D, Tognoni G, Defilippi G, Buccheri D, Tespili M, Corrado D, Steffenino G; BVS-RAI investigators. Registro Absorb Italiano (BVS-RAI): an investigators-owned and -directed, open, prospective registry of consecutive patients treated with the Absorb BVS: study design. Cardiovasc Revasc Med. 2015 Sep;16(6):340-3. doi: 10.1016/j.carrev.2015.05.010. Epub 2015 Jun 3. PMID 26100975